CLINICAL TRIAL: NCT03959475
Title: A Descriptive Multicenter Investigation of Geriatrics Hotlines : Description of the Health Care Pathways and Conditions of Subjects Aged 75 and Over
Brief Title: A Descriptive Multicenter Investigation of Geriatrics Hotlines : A French Study
Status: Completed | Type: Observational
Sponsor: Support and Education Technic Centre (Other)
Collaborators: National School for Social Security (Unknown); Loire department (Unknown)
Responsible Party: Principal Investigator, Régis Gonthier, Profesor, Centre Hospitalier Universitaire de Saint Etienne
Other Study IDs: CFPPA-Loire-Hotline-2018
Record Dates: First submitted 2019-05-16; First posted 2019-05-22 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Geriatric; Elderly
Keywords: Elderly subject; healthcare; Hotline; emergency department; GP medicine
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Saint-Etienne Hospital: All people aged 75 years and over hospitalized in short-stay geriatric care via a hotline in this hospital
- Firminy hospital: All people aged 75 years and over hospitalized in short-stay geriatric care via a hotline in this hospital
- South Lyon hospital: All people aged 75 years and over hospitalized in short-stay geriatric care via a hotline in this hospital
- Bordeaux hospital: All people aged 75 years and over hospitalized in short-stay geriatric care via a hotline in this hospital
- Saint-Chamond hospital: All people aged 75 years and over hospitalized in short-stay geriatric care via a hotline in this hospital
- Angers hospital: All people aged 75 years and over hospitalized in short-stay geriatric care via a hotline in this hospital
- Clermont Ferrand hospital: All people aged 75 years and over hospitalized in short-stay geriatric care via a hotline in this hospital

SUMMARY:
In France, for general practitioners, the Emergency Hospitality Services (UAS) are the fastest and usual way to respond to the complexity of managing elderly polypathological patients. In 2013, the Regional Health Agencies proposed the creation of direct telephone assistance managed by geriatric doctors (geriatric hotlines) to promote interactions city - hospital. The aim of these hotlines is to improve the care pathways and health status of seniors. The objective of this study is to describe the care trajectories and health status of subjects over 75 years of age hospitalized in a short-term geriatric stay on the guidance of a Geriatric Hotline.

The study will take place over 24 months and in 7 French University Hospitallers Centres. The study will include all patients aged 75 and over, living at home or in an institution, who are hospitalized in a short-term geriatric ward on the guidance of a Hotline.

The results will show whether a management by the geriatric hotline is the most suitable for seniors, with an average length of stay probably shorter.

DETAILED DESCRIPTION:
This is a multicenter descriptive study conducted in seven French investigating centers (including university centers) with sub-group analysis. Participating establishments will all be voluntary. In order to participate to the study, an establishment must have a specific telephone line for doctor-doctor communications. Only calls originating from healthcare professionals are to be taken into account.

The study will last for 24 months. Study population and eligibility The study population will be constituted of people aged 75 and over, living in their own home or in a care facility (including independent-living facilities), hospitalized in short-stay geriatric care referred by the hotline in one of the investigating centers, and who are fully aware of the study and their rights regarding their participation. The first questionnaire will be filled out via the hotline by the geriatric specialist answering the call. A second questionnaire will then be filled out during the patient's hospitalization by the treating geriatric specialist

Recruitment:

All people aged 75 years and over hospitalized in short-stay geriatric care via a hotline.

Inclusion:

Inclusion procedure: (the location, inclusion and non-inclusion criteria verification by investigators, explanation of the study, and delivery of information form will all be the responsibility of each center independently, conducted when the patient is admitted to short-stay geriatric care).

Monitoring:

This study involves no extra examinations or treatment besides traditional practices, the only difference being the digitization of all medical findings for analysis.

Study endpoint:

This corresponds to when the patient is discharged from short-stay geriatric care.

Study participation duration for each patient: short-stay geriatric care duration.

SELECTION AND EXCLUSION OF SUBJECTS FROM STUDY Inclusion criteria

* Age ≥75 years
* Male/Female
* Living in own home or in a care facility (including independent-living facilities)
* Hospitalized in short-stay geriatric care
* Confirmed receipt of information on the study and their rights, as stipulated by articles L. 1122-1 of the French public health code, by 57 of the "Informatique et Libertés" data protection act, and by MR-003 of the French data protection and civil liberties authority (CNIL).

Non-inclusion criteria for people seeking participation

* Patients less than 75 years of age
* Refusal to participate

Procedure for early discontinuation of the study or exclusion from the study All subjects can, at any moment and by any method, decide to withdraw from the study.

Evaluation criteria The primary endpoint is the mean duration of hospitalization in short-stay geriatric care.

The secondary endpoints selected are hospital mortality rate, assessment of health status of elderly patients hospitalized in short-stay geriatric wards using different criteria, and their outcomes following discharge; describing and comparing how the different hotlines across France function; analyzing the principal responses provided to doctors using the hotline and improving awareness.

This study will be noninterventional. All interventions will be carried out following normal clinical practices. There will be no unusual risk or specific constraint for participating patients.

RECORDED VARIABLES AND SOURCE DATA The study data will be collected directly from the questionnaires as the study progresses.

For the first questionnaire, filled out by the hotline geriatric specialist, the following information will be collected for the study:

Health data: the identification of both speakers on the call; patient age; reasons for calling; degree of emergency as perceived by the geriatric specialist and the calling doctor, evaluated by simple verbal scale from 0 to 10; responses offered by geriatric specialist.

Administrative data: call duration in minutes. This questionnaire will be anonymous with no identifying criteria. It will be filled out every time contact is made via the hotline, irrespective of what responses are offered by the doctor (referrals to short-stay geriatric care or not).

For the second questionnaire, filled out by the geriatric specialist treating the patient during their hospitalization in short-stay geriatric care, following referral from the hotline, the following information will be collected for the study:

Socio-demographic data: First and last name of the patient, Patient Permanent Identification (PPI) number, patient age. This data will be anonymized on entry.

Health data: Reasons for hospitalization, number of hospitalizations during the year, polypharmacy (>4), biological data : albumin and C-reactive protein levels for assessing nutritional status, Charlson's index calculation using patient history for assessing the comorbidities of our geriatric population), evaluation of activities of daily living (ADL) prior to hospitalization according to the validated ADL (/6) and instrumental ADL (IADL) scales (/4), evaluation of cognitive status using MMSE score (/30), recommended referral after hospital discharge.

Family/Marital status data: single or with a partner, with or without children Living situation data: Residence of patient (own home, independent-living facility, nursing home) Type of living area data: urban, semi-urban or rural

Signaling data and findings relating to family or marital status will help characterize the patients who participate.

Data relating to living location, type and area are recorded in order to assess the impact of these factors on use of the hotline.

Finally, data relating to health status is recorded as justified by the bibliographical references to which it is sent.

ELIGIBILITY:
Inclusion Criteria:

* Age over 75
* Male/Female
* Living at home or in an institution (independent residence included)
* Being hospitalized in a short geriatric stay

Exclusion Criteria:

* Patients under 75 years
* Refusal to participate in study

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population will be constituted of people aged 75 and over, living in their own home or in a care facility (including independent-living facilities), hospitalized in short-stay geriatric care referred by the hotline in one of the investigating centers, and who are fully aware of the study and their rights regarding their participation.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2018-05-05 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
the mean duration of hospitalization in short-stay geriatric care | through study completion, an average of 2 years
  the mean duration of hospitalization in short-stay geriatric care

SECONDARY OUTCOMES:
Assessment of health status using the Charlson comorbidity index for elderly patients hospitalized in short-stay geriatric wards | through study completion, an average of 2 years
  By questionnaire : Charlson's index calculation using patient history for assessing the comorbidities of our geriatric population.
  The Charlson comorbidity index : a method of predicting mortality by classifying or weighting comorbid conditions.
  The Charlson comorbidity index predicts the one-year mortality for a patient who may have a range of comorbid conditions, such as heart disease, AIDS, or cancer (a total of 22 conditions). Each condition is assigned a score of 1, 2, 3, or 6, depending on the risk of dying associated with each one. Scores are summed to provide a total score to predict mortality The minimum score is 0 and the maximum score is 27. The value 0 is the best possible result. With a charlson score of 3 or higher, there is a risk of an adverse change in the patient's state of health.
  Score = 0 => 12% of 1 year mortality Score of 1 to 2 => 26% of 1 year mortality Score of 3 to 4 => 52% of 1 year mortality Score of 5 or more => 85% of 1 year mortality
Describing and comparing how the different hotlines across France function | through study completion, an average of 2 years
  By questionnaire for all hotlines : N° residents, total number of hospital beds, short-stay geriatric care Yes/No, post-discharge care Yes/No, long-term rehabilitation care Yes/No, consultation Yes/No, Outpatient clinic Yes/No, Ambulance care Yes/No, telemedical consultation Yes/No.

CONTACTS AND LOCATIONS:
Overall Officials: Régis GONTHIER, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

REFERENCES:
- [Derived] Mourgues C, Bongue B, Dupre C, Goethals L, Celarier T, Blanquet M. Geriatric Helpline Services to Improve Health and Care Pathways in Older Adults: A Cost-Effectiveness Analysis. Health Sci Rep. 2025 Dec 8;8(12):e71635. doi: 10.1002/hsr2.71635. eCollection 2025 Dec. PMID 41377772
- [Derived] Goethals L, Barth N, Martinez L, Lacour N, Tardy M, Bohatier J, Bonnefoy M, Annweiler C, Dupre C, Bongue B, Celarier T. Decreasing hospitalizations through geriatric hotlines: a prospective French multicenter study of people aged 75 and above. BMC Geriatr. 2023 Nov 28;23(1):783. doi: 10.1186/s12877-023-04495-9. PMID 38017388
- [Derived] Martinez L, Lacour N, Gonthier R, Bonnefoy M, Goethals L, Annweiler C, Salles N, Jomard N, Bohatier J, Tardy M, Ojardias E, Jugand R, Bongue B, Celarier T. Impact of Geriatric Hotlines on Health Care Pathways and Health Status in Patients Aged 75 Years and Older: Protocol for a French Multicenter Observational Study. JMIR Res Protoc. 2020 Feb 13;9(2):e15423. doi: 10.2196/15423. PMID 32053116